CLINICAL TRIAL: NCT04906707
Title: Home-Based Intervention for Chronic Pain in Adults With Sickle Cell Disease (HIPAS)
Brief Title: Home-Based Intervention for Chronic Pain in Adults With Sickle Cell Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Nadine Matthie, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00002004; 1R21NR019872-01 (NIH)
Record Dates: First submitted 2021-05-27; First posted 2021-05-28 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Sickle Cell Disease
Keywords: Pain management; Virtual Reality Device
MeSH Terms: conditions — Anemia, Sickle Cell; Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- EaseVRx Group (Experimental): Participants will be asked to complete the 8-week program with assigned modules each week. Each week, participants will be asked to complete 7 modules, averaging 5 minutes in duration and ranging from 2 to 16 minutes in duration, for a total of 56 modules across the program. Participants will be instructed not to use the device while ambulating, and that they should use the headset a maximum of 3 times per 24-hour period (morning, noon, and evening) for not more than 30 minutes consecutively.
  Interventions: Device: EaseVRx
- Active control Group (Active Comparator): Participants in the control group will be asked to use the audio-only version of EaseVRx that excludes references to visual content. They will receive an electronic link to the audio recordings on SoundCloud (a music streaming platform) where they can choose to stream or download the audio recordings on their smartphone, laptop, or desktop computer. Each week, participants will be asked to complete 7 audio sessions.
  Interventions: Behavioral: Audio-only version of EaseVRx

INTERVENTIONS:
Device: EaseVRx — EaseVRx is a commercially available pain management program. It is a multi-modal, skills-based, 8-week, VR, mind-body approach to daily management of chronic pain that is designed for home use to be worn over the eyes. The program contains five types of modules that are as follows: Interoception, Education, 360-degree relaxation videos, Games, and Dynamic breathing. All program content is mapped to a therapeutically designed curriculum with weekly themes. The following core themes are infused into the curriculum: Acceptance, Attention shifting, Awareness, Rehabilitation, Self-compassion, Healthy Movement, Deep relaxation, Visualization, Knowledge of pain, Distraction, and Immersive enjoyment.
  Arms: EaseVRx Group
Behavioral: Audio-only version of EaseVRx — Participants in the control group will be asked to use the audio-only version of EaseVRx, which excludes references to visual content, to complete 7 sessions weekly. They will receive an electronic link to the recordings on SoundCloud (a music streaming platform) where they can choose to stream or download the audio recordings on their smartphone, laptop, or desktop computer.
  Arms: Active control Group

SUMMARY:
This project will evaluate AppliedVR's EaseVRx - a multi-modal, skills-based, 8-week, virtual reality, home intervention - in an exploratory randomized controlled trial for self-management of chronic pain among Black, young adults (ages 18-50) with sickle cell disease.

DETAILED DESCRIPTION:
Chronic pain in sickle cell disease (SCD) is a major health problem. Because of the high pain burden associated with SCD and the existing health disparities in comprehensive pain management, non-pharmacological, home-based strategies are urgently needed to help manage chronic pain. In this study, the investigators will use a single-site, 8-week, randomized clinical trial (with follow-up at 12 weeks) to evaluate a home-based, pain self-management program for chronic pain in Black adults with SCD. Study participants will be identified from the group of patients with chronic pain who receive care in the SCD clinic of the Georgia Comprehensive Sickle Cell Center at Grady Memorial Hospital (Grady) in Atlanta, Georgia. Patients may be recommended by the Center's staff or may self-identify in response to study flyers posted in the Center, health facilities or community-based organizations in surrounding areas, or on social media. Recruitment and consent will take place in a private area of the SCD clinic, the research center in the Nell Hodgson Woodruff School of Nursing at Emory University, or remotely if necessary. Consent may also occur remotely if necessary.

After enrollment, in-person study activities will take place in the SCD clinic or the research center while remote study activities will take place in participants' homes on their own time. Participants will complete questionnaires and a pain diary, use the pain management program at home (delivered with a virtual reality device or audio only on SoundCloud), and complete a qualitative interview or focus group session. Compensation will be provided after completion of each of these study activities. During the study, subjects will continue their standard pain management routine, including any pain medications, as prescribed by their healthcare provider.

This research will advance both scientific knowledge and human health by focusing on addressing unmet needs for an underserved population. This study is the first randomized clinical trial that investigates a virtual reality, home-based pain self-management program for chronic pain in adults with SCD. Therefore, this study represents the first essential step in developing a culturally-tailored, non-pharmacological, home-based, chronic pain self-management intervention specifically for Black adults with SCD that can be used along with standard SCD care.

ELIGIBILITY:
Inclusion Criteria:

* Black adults,
* ages 18-50 years;
* diagnosis of SCD (Sickle cell disease);
* chronic non vaso-occlusive pain experienced > 3 days per week on average for > 6 months;
* ability to wear a VR (Virtual reality) head-mounted display and move head in cervical rotation, extension, and flexion; sufficient fine motor control to operate VR equipment such as a controller; and ability to read, write, and understand English.

Exclusion Criteria:

* 1. Conditions: Co-morbidities that may influence pain perception; diagnosis of epilepsy or susceptibility to seizures, migraines, or other neurological disorders that may prevent VR use, and/or other medical conditions due to which individuals are predisposed to nausea and dizziness; susceptibility to claustrophobia, motion sickness or cybersickness (digital motion sickness); history of blackouts; hypersensitivity to flashing lights or motion; lack of stereoscopic vision; severe visual or hearing impairment; inability to operate VR equipment (such as inability to turn head or use hands to operate external controller); and/or injury to the eyes, face, head, or neck that prevents comfortable VR use.

  2. Other exclusions: Medical instability as determined by healthcare providers at the study site; significant motor impairment; surgery within the last three months; planning to start a new pain management strategy (such as medication, physiotherapy, acupuncture, or cognitive behavioral therapy) in the next three months; history of major psychiatric disorder (such as schizophrenia or bipolar disorder) not controlled with medication or behavioral factors that would interfere with study procedures; alcohol or substance dependence, heart conditions, or the presence of implanted medical devices (such as cardiac pacemakers) as noted in the electronic health record; cognitive or developmental disabilities; active suicidal ideation; inability to read, write, or understand English; pregnancy; and/or plans for vacation in the next three months.

This study will not include any of these special populations:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Matthie, PhD, RN, CNL, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital - Outpatient Sickle Cell Clinic, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
* Individual participant data that underlie the results reported, after de-identification (text, tables, figures, and appendices)
  * Investigators whose proposed used of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose
  * For individual participant data meta-analysis
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Proposals may be submitted up to 36 months following article publication. After 36 months, the data will be available in our University's data warehouse but without investigator support other than deposited metadata.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EaseVRx Group | Active Control Group
Started | 19 | 25
Completed | 16 | 24
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Withdrawal due to PI decision | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EaseVRx Group | Active Control Group | Total
Number analyzed (Participants) | 19 | 25 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.37 (6.67) | 31.72 (7.61) | 33.73 (7.50)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 7 | 9 | 16
  Transgender Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 19 | 23 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 24 | 41
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 19 | 25 | 44

OUTCOME MEASURES:

1. Primary Outcome: Pain Rating Using Numerical Pain Rating Scale (NPRS)
Description: For daily measures, self-reported pain ratings will be assessed with the Numerical Pain Rating Scale (NPRS). On the NPRS, pain intensity levels range from 0 to 10 (0 = no pain and 10 = worst pain). Lower pain ratings correlate with better outcome.
  Daily Pain Diary responses were intermittent and can only be aggregated during time period 1 (days 1-28) and time period 2 (days 29-56). Diaries were not administered at day 0.
Time Frame: Baseline, up to week 4 or time period 1 (day 1-28), from week 4 to 8 or time period 2 (days 29-56)
Population: Participants who completed the corresponding survey for this outcome are included per timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 12 | 23
score on a scale
  NPRS daily score at up to week 4 or time period 1 (day 1-28) | 3.79 (2.93) | 3.17 (2.79)
  NPRS daily score from week 4 to 8, or time period 2 (days 29-56) | 2.37 (2.77) | 2.63 (2.78)

2. Primary Outcome: Pain Intensity Subscale of the Chronic Pain Grade Questionnaire
Description: For baseline and monthly measurements, self-reported pain ratings were assessed with the Pain Intensity subscale of the Chronic Pain Grade Questionnaire. On the Chronic Pain Grade Questionnaire, pain intensity levels range from 0-100. Lower pain ratings correlate with better outcome.
Time Frame: Baseline, week 4, week 8, and 4 weeks post-intervention (week 12)
Population: Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 19 | 25
score on a scale
  Pain Intensity score at Baseline | 66.84 (12.64) | 63.07 (15.84)
  Pain Intensity score at 4 weeks: number analyzed (Participants) | 12 | 23
  Pain Intensity score at 4 weeks | 60.28 (13.06) | 54.06 (16.24)
  Pain Intensity score at 8 weeks: number analyzed (Participants) | 10 | 23
  Pain Intensity score at 8 weeks | 56.33 (13.65) | 48.84 (17.68)
  Pain Intensity score at 12 weeks: number analyzed (Participants) | 10 | 19
  Pain Intensity score at 12 weeks | 60.00 (14.05) | 45.96 (20.54)

3. Primary Outcome: Participant Engagement: Minutes of Program Use Per Day
Description: Minutes of daily program use may range from 2 minutes to 48 minutes or more. The investigator hypothesizes that higher usage will correlate with a better outcome.
  Because of intermittent usage patterns, self-reported program use was aggregated during time period 1 (days 1-28) and time period 2 (days 29-56).
Time Frame: up to week 4 or time period 1 (day 1-28), from week 4 to 8 or time period 2 (days 29-56)
Population: Participants who completed the corresponding survey for this outcome are included per timepoint
Measure: Median (Inter-Quartile Range); unit: Minutes of Program Use Per Day
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 19 | 24
Minutes of Program Use Per Day
  Time period 1 (days 1-28) | 170.5 [18.75 to 314.0] | 128.5 [56.25 to 197.44]
  Time period 2 (days 29-56): number analyzed (Participants) | 16 | 24
  Time period 2 (days 29-56) | 243.0 [18.75 to 477.5] | 163.25 [66.25 to 315.85]

4. Primary Outcome: Participant Engagement: Duration in Days
Description: Throughout the 8-week treatment period, device usage duration may range from 0 to 7 days each week. The investigator hypothesizes that higher usage will correlate with a better outcome.
Time Frame: Baseline, daily during treatment (4 weeks or time period 1, day 1-28), daily during treatment (8 weeks or time period 2, days 29-56)
Population: Lack of granularity in the VR device usage data (data provided monthly, not daily) limits the ability to identify specific usage patterns for reporting regarding duration in minutes each week. However, usage duration was self-reported by the VR group and the audio group. Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 18 | 23
days
  Time period 1 (days 1-28) | 1.38 [0.25 to 3.33] | 2.75 [1.5 to 5.3]
  Time period 2 (days 29-56): number analyzed (Participants) | 14 | 22
  Time period 2 (days 29-56) | 1.63 [0.20 to 4.2] | 2.13 [0.95 to 4.13]

5. Primary Outcome: Participant Engagement: Features Utilized
Description: Assessed by the number of features utilized when using the VRdevice. The number of features utilized may be 1 or 2 . The investigator hypothesizes that use of a higher number of features will correlate with a better outcome.
Time Frame: Daily during treatment (8 weeks)
Population: Lack of granularity in the VR usage data limits the ability to identify specific usage patterns. Therefore, the average number of features utilized can only be reported across the 8 weeks of treatment. Participants who completed the corresponding survey for this outcome are included per timepoint.
  This outcome was not applicable to the Audio group.
Measure: Count of Participants; unit: Participants
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 17 | 0
Participants
  Number of participants with 1 feature utilized | 6 |
  Number of participants with 2 features utilized | 11 |

6. Primary Outcome: Participant Engagement: Completion Rates
Description: Assessed by completion rates: the number of modules completed weekly. Rates may range from 0 to 7 modules completed each week. The investigator hypothesizes that completion of a higher number of modules weekly will correlate with a better outcome.
Time Frame: Daily average during treatment (up to 8 weeks)
Population: Because of intermittent usage patterns, the average number of modules completed weekly could not be assessed for the Audio group (Active control group).
  Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Mean (Inter-Quartile Range); unit: modules/week
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 16 | 0
modules/week | 2.38 [0.44 to 5.01] |

7. Primary Outcome: Study Retention: Surveys
Description: Assessed by participant completion of survey measures at repeated timepoints (baseline, week 4, week 8, and week 12). The investigator hypothesizes that higher study retention will correlate with a better outcome.
Time Frame: Baseline, 4 weeks, 8 weeks and 4 weeks post-intervention (week 12)
Population: Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Number; unit: surveys completed
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 19 | 25
surveys completed
  Baseline | 19 | 25
  4 weeks | 12 | 23
  8 weeks | 10 | 23
  4 weeks post-intervention (week 12) | 10 | 19

8. Primary Outcome: Study Retention: Daily Diaries
Description: Assessed by participant completion of daily diaries across 8 weeks of treatment (days 1-56). The investigator hypothesizes that higher study retention will correlate with a better outcome.
Time Frame: Up to 8 weeks
Population: Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Number; unit: daily diaries
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 18 | 24
daily diaries | 28 | 32

9. Primary Outcome: Participant Satisfaction
Description: Assessed, once at the end of the program, via individual qualitative interviews or focus group sessions. Participants will be asked to evaluate the program by responding to the four items listed below, using a Likert scale (strongly agree, somewhat agree, somewhat disagree, strongly disagree with possible score range 1-4) for the first three items and 1-10 (with 10 being definitely would recommend) for the fourth item.• The VR program was easy to use.• I enjoyed using the VR program.• The content in the VR program helped me cope with my pain.• On a scale of 1-10, how likely are you to recommend the VR program to someone else at this time? The investigator hypothesizes that responses of strongly agree and higher scores will correlate with a better outcome.
Time Frame: Post-treatment (up to 6 weeks post-treatment)
Population: Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 8 | 16
score on a scale
  The program was easy to use (Scale of 1-4) | 4.0 [3.0 to 4.0] | 4.0 [3.0 to 4.0]
  I enjoyed using the program (Scale of 1-4) | 4.0 [3.0 to 4.0] | 4.0 [3.0 to 4.0]
  The content in the program helped me cope with my pain (Scale of 1-4) | 4.0 [3.0 to 4.0] | 4.0 [3.0 to 4.0]
  On a scale of 1-10, how likely are you to recommend the program to someone else at this time? | 10.0 [7.0 to 10.0] | 10.0 [8.0 to 10.0]

10. Primary Outcome: Frequency of Highest Satisfaction Scores
Description: Assessed once at the end of the program, via individual qualitative interviews or focus group sessions.
  Participants choosing the highest score for each of the four items listed will be counted.
  Higher number correlates with a better outcome.
Time Frame: Post-treatment (up to 6 weeks post-treatment)
Population: Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 8 | 16
Participants
  Participants with highest score for "The program was easy to use" | 7 | 14
  Participants with highest score for "I enjoyed using the program" | 6 | 13
  Participants with highest score for "The content in the program helped me cope with my pain" | 6 | 12
  Participants with highest score for "how likely you to recommend the program to someone else?" | 5 | 9

11. Primary Outcome: Safety: Number of Adverse Events
Description: Assessed by monitoring participants for the number of adverse events. Fewer adverse events correlate with a better outcome.
Time Frame: 4 weeks, 8 weeks, up to 6 weeks post-treatment
Population: This outcome was only assessed in the EaseVRx Group because it was not applicable to the Audio group .Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Number; unit: adverse events
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 16 | 0
adverse events
  Number of Adverse events at 4 weeks | 2 |
  Number of Adverse events at 8 weeks | 0 |
  Number of adverse events at up to 6 weeks post-treatment | 0 |

12. Secondary Outcome: Chronic Pain Acceptance Score
Description: Assessed by the Chronic Pain Acceptance Questionnaire (CPAQ-8) which measures acceptance of chronic pain. Items are scored on a scale from 0 to 6 (never true to always true), and higher scores (total possible scores range from 0 to 48) indicate higher levels of acceptance (better outcome).
Time Frame: Baseline, week 4, week 8 and 4 weeks post-intervention (week 12)
Population: Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 19 | 25
score on a scale
  Baseline | 24.00 (7.83) | 21.40 (5.97)
  Week 4: number analyzed (Participants) | 11 | 23
  Week 4 | 26.45 (6.99) | 23.43 (4.80)
  Week 8: number analyzed (Participants) | 10 | 23
  Week 8 | 28.20 (5.90) | 23.65 (6.73)
  Week 12: number analyzed (Participants) | 10 | 19
  Week 12 | 28.30 (5.02) | 25.26 (3.45)

13. Secondary Outcome: Chronic Pain Self-Efficacy
Description: Assessed by using the Chronic Pain Self-Efficacy Scale (CPSES), which measures efficacy expectations for coping with the consequences of chronic pain. Items are scored on a 10-point Likert-type scale from 1 (very uncertain) to 10 (very certain), with a minimum total score of 22 and a maximum total score of 220. Higher scores indicate a better outcome.
Time Frame: Baseline, week 4, week 8, and 4 weeks post-intervention (Week 12)
Population: Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 19 | 25
score on a scale
  Baseline | 154.68 (27.70) | 155.92 (32.60)
  Week 4: number analyzed (Participants) | 11 | 23
  Week 4 | 155.82 (42.36) | 151.52 (35.25)
  Week 8: number analyzed (Participants) | 10 | 23
  Week 8 | 166.40 (31.01) | 148.13 (42.82)
  Week 12: number analyzed (Participants) | 10 | 19
  Week 12 | 162.60 (24.93) | 160.89 (39.33)

14. Secondary Outcome: Social Support
Description: Assessed by using the Social Support Questionnaire (SSQ), which measures perceptions of the desirability, availability, use, and usefulness of social support. Items are scored on a scale from 1 (not at all) to 5 (very much, constantly), with a minimum total score of 32 and a maximum total score of 160. Higher scores indicate a better outcome.
Time Frame: Baseline, week 4, week 8, and 4 weeks post-intervention (12 weeks)
Population: Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 19 | 25
score on a scale
  Baseline SSQ score | 111.95 (23.81) | 123.48 (24.57)
  Week 4 SSQ score: number analyzed (Participants) | 11 | 23
  Week 4 SSQ score | 116.55 (27.26) | 129.48 (18.78)
  Week 8 SSQ score: number analyzed (Participants) | 10 | 25
  Week 8 SSQ score | 115.50 (33.37) | 121.52 (22.78)
  Week 12 SSQ score: number analyzed (Participants) | 10 | 19
  Week 12 SSQ score | 121.90 (19.94) | 131.89 (23.02)

15. Secondary Outcome: Pain Catastrophizing Score
Description: Assessed by using the Pain Catastrophizing Scale (PCS-13) which measures thoughts and feelings when pain is experienced. Items are scored on a scale from 0 to 4 (not at all to all the time), and higher scores (scores range from 0 to 52) indicate a higher degree of catastrophizing (worse outcome).
Time Frame: Baseline, week 4, week 8 and 4 weeks post-intervention (week 12)
Population: Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 19 | 25
score on a scale
  Baseline | 22.74 (14.80) | 25.48 (10.78)
  Week 4: number analyzed (Participants) | 11 | 23
  Week 4 | 18.82 (8.20) | 21.91 (11.80)
  Week 8: number analyzed (Participants) | 10 | 23
  Week 8 | 14.30 (7.10) | 19.26 (9.63)
  Week 12: number analyzed (Participants) | 10 | 19
  Week 12 | 14.50 (5.80) | 18.00 (11.35)

16. Secondary Outcome: BRIEF Health Literacy Score
Description: Assessed by using the BRIEF Health Literacy Screening Tool which measures the amount of help needed in healthcare situations. Items are scored on a scale from 1 to 5 (always to never and not at all to extremely), and higher total scores (scores range from 4 to 20) indicate greater health literacy (better outcome).
Time Frame: Baseline, week 4, week 8, and 4 weeks post-intervention (Week 12)
Population: Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 19 | 25
score on a scale
  Baseline | 19.05 (1.39) | 18.24 (2.33)
  Week 4: number analyzed (Participants) | 12 | 23
  Week 4 | 19.00 (1.79) | 17.65 (3.01)
  Week 8: number analyzed (Participants) | 10 | 23
  Week 8 | 18.60 (2.37) | 17.04 (3.01)
  Week 12: number analyzed (Participants) | 10 | 19
  Week 12 | 19.00 (1.89) | 17.84 (2.99)

17. Secondary Outcome: Executive Function
Description: Behavior Rating Inventory of Executive Function (BRIEF-A) which measures adult executive functioning/self-regulation. Items are scored on a scale from 1 to 7 (never a problem to always a problem) and higher total scores (scores range from 34 to 238) indicate more symptoms of executive dysfunction (worse outcome).
Time Frame: Baseline, week 4, week 8, and 4 weeks post-intervention (week 12)
Population: Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 19 | 25
score on a scale
  Baseline BRIEF-A score | 78.53 (24.02) | 98.12 (28.50)
  BRIEF-A score at Week 4: number analyzed (Participants) | 11 | 23
  BRIEF-A score at Week 4 | 76.27 (26.41) | 83.00 (25.71)
  BRIEF-A score at Week 8: number analyzed (Participants) | 10 | 23
  BRIEF-A score at Week 8 | 79.00 (25.83) | 92.43 (28.80)
  BRIEF-A score at Week 12: number analyzed (Participants) | 10 | 19
  BRIEF-A score at Week 12 | 75.90 (17.65) | 79.74 (28.17)

18. Secondary Outcome: Anxiety Levels
Description: Assessed by using PROMIS Emotional Distress - Anxiety (Anxiety 8a - Adult v1.0), which measures self-reported fear, anxious misery, hyperarousal, and somatic symptoms related to arousal. Items are scored on a 5-point Likert scale ranging from 1 (never) to 5 (always) and the total raw score (minimum total score of 8 and maximum total score of 40) is rescaled into a standardized T-score. The standardized T-score, with a minimum total score of 37.1 and a maximum total score of 83.1, has a mean of 50 and a standard deviation of 10. Higher T-scores indicate a worse outcome.
Time Frame: Baseline, week 4, week 8 and 4 weeks post-intervention (week 12)
Population: Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 19 | 25
T-score
  Baseline | 53.19 (9.33) | 57.38 (8.43)
  Week 4: number analyzed (Participants) | 11 | 23
  Week 4 | 52.65 (10.21) | 56.74 (9.70)
  Week 8: number analyzed (Participants) | 10 | 23
  Week 8 | 47.72 (8.45) | 54.65 (8.85)
  Week 12: number analyzed (Participants) | 10 | 19
  Week 12 | 50.03 (11.14) | 52.56 (10.83)

19. Secondary Outcome: Depression Levels
Description: Assessed by using PROMIS Emotional Distress - Depression (Depression 8a - Adult v1.0), which measures self-reported negative mood, views of self, social cognition, and decreased positive affect and engagement. Items are scored on a 5-point Likert scale ranging from 1 (never) to 5 (always) and the total raw score (minimum total score of 8 and maximum total score of 40) is rescaled into a standardized T-score. The standardized T-score, with a minimum total score of 38.2 and a maximum total score of 81.3, has a mean of 50 and a standard deviation of 10. Higher T-scores indicate a worse outcome.
Time Frame: Baseline, week 4, week 8 and 4 weeks post-intervention (week 12)
Population: Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 19 | 25
T-score
  Baseline | 48.96 (8.66) | 55.60 (10.03)
  Week 4: number analyzed (Participants) | 11 | 23
  Week 4 | 48.59 (7.78) | 53.50 (9.97)
  Week 8: number analyzed (Participants) | 10 | 23
  Week 8 | 45.99 (9.71) | 52.94 (8.81)
  Week 12: number analyzed (Participants) | 10 | 19
  Week 12 | 45.05 (8.71) | 49.15 (9.56)

20. Secondary Outcome: Sleep Impact Short Form Score
Description: Assessed by using the Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-Me) Sleep Impact Short Form, which measures sleep disturbances. 5 items are assessed using a scale that ranges from 1 (never or always) to 5 (never or always) and the total raw score (minimum total score of 5 and maximum total score of 25) is rescaled into a standardized T-score. The standardized T-score, with a minimum total score of 27.9 and a maximum total score of 69.1, has a mean of 50 and a standard deviation of 10. Higher T-scores indicate a better outcome.
Time Frame: Baseline, week 4, week 8 and 4 weeks post-intervention (week 12)
Population: Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 19 | 25
T-score
  Baseline | 49.03 (7.04) | 49.92 (5.48)
  Week 4: number analyzed (Participants) | 11 | 23
  Week 4 | 49.75 (7.56) | 50.65 (6.20)
  Week 8: number analyzed (Participants) | 10 | 23
  Week 8 | 52.91 (5.68) | 51.64 (5.91)
  Week 12: number analyzed (Participants) | 10 | 19
  Week 12 | 55.37 (6.15) | 51.88 (7.17)

21. Secondary Outcome: Functional Activities of Daily Living
Description: Assessed by using the Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-Me) Pain Impact Short Form, which measures the effects of sickle cell pain on activities of daily living. 5 items are assessed using a scale that ranges from 1 (always) to 5 (never) and the total raw score (minimum total score of 5 and maximum total score of 25) is rescaled into a standardized T-score. The standardized T-score, with a minimum total score of 24.8 and a maximum total score of 63.8, has a mean of 50 and a standard deviation of 10. Higher T-scores indicate a better outcome.
Time Frame: Baseline, week 4, week 8 and 4 weeks post-intervention (week 12)
Population: Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 19 | 25
T-score
  Baseline | 49.65 (6.39) | 47.81 (6.68)
  Week 4: number analyzed (Participants) | 11 | 23
  Week 4 | 51.77 (7.07) | 47.30 (6.66)
  Week 8: number analyzed (Participants) | 10 | 23
  Week 8 | 51.54 (6.86) | 48.06 (8.43)
  Week 12: number analyzed (Participants) | 10 | 19
  Week 12 | 52.59 (8.62) | 49.44 (9.78)

22. Secondary Outcome: Chronic Pain Disability Score
Description: Assessed by the Chronic Pain Grade Questionnaire (CPGQ) which classifies individuals into one of four categories according to pain severity or interference. Items are scored on a scale from 0 to 10, with total scores for chronic pain intensity and chronic pain disability ranging from 0 to 100. Higher total scores indicate a higher level of disability that is severely limiting (worse outcome).
Time Frame: Baseline, week 4, week 8, and 4 weeks post-intervention (week 12)
Population: Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 19 | 25
score on a scale
  Baseline | 56.14 (26.42) | 54.67 (24.29)
  Week 4: number analyzed (Participants) | 12 | 23
  Week 4 | 48.06 (21.67) | 51.01 (20.68)
  Week 8: number analyzed (Participants) | 10 | 23
  Week 8 | 39.33 (17.90) | 44.20 (17.06)
  Week 12: number analyzed (Participants) | 10 | 19
  Week 12 | 43.00 (14.61) | 42.81 (27.45)

23. Secondary Outcome: Average Healthcare Utilization
Description: Assessed by healthcare utilization for pain in the previous 12 months as reflected by self-reported number of healthcare visits. The number of healthcare visits may range from 0 to 20 or more. A higher number of visits is correlated with worse outcome.
Time Frame: Baseline
Population: Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Median (Inter-Quartile Range); unit: healthcare visits
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 22 | 25
healthcare visits | 2.5 [0.0 to 5.0] | 2.0 [1.0 to 5.5]

24. Secondary Outcome: Number of Analgesics
Description: Assessed by self-reported number of over-the-counter analgesics used per day via the Daily Pain Diary. Results will be reported during time period 1 (days 1-28) and time period 2 (days 29-56). A higher number of pain medications correlates with a worse outcome.
Time Frame: Time period 1 (days 1-28) and time period 2 (days 29-56)
Population: Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Mean (Standard Deviation); unit: analgesics/day
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 19 | 25
analgesics/day
  Time period 1 (days 1-28) | 4.88 (3.35) | 3.80 (3.01)
  Time period 2 (days 29-56) | 4.86 (2.18) | 4.69 (3.64)

25. Secondary Outcome: Quality of Life: Frequency of Sickle Cell Pain Episodes
Description: Assessed by using the Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-Me) Pain Episodes Short Form, which measures the frequency and severity of sickle cell pain episodes. 2 items are assessed using a scale that varies across the items, with values ranging from 0-4 or 0-7, and the total raw score (minimum total score of 0 and maximum total score of 11) is rescaled into a standardized T-score. The standardized T-score has a mean of 50 and a standard deviation of 10. Higher T-scores indicate a worse outcome.
Time Frame: Baseline, week 4, week 8, and 4 weeks post-intervention (week 12)
Population: Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 19 | 25
T-score
  Baseline | 51.85 (8.39) | 47.65 (8.97)
  Week 4: number analyzed (Participants) | 11 | 23
  Week 4 | 50.08 (8.22) | 46.27 (11.88)
  Week 8: number analyzed (Participants) | 10 | 23
  Week 8 | 48.74 (10.81) | 45.93 (12.83)
  Week 12: number analyzed (Participants) | 10 | 19
  Week 12 | 47.96 (9.69) | 42.23 (12.58)

26. Secondary Outcome: Quality of Life: Severity of Sickle Cell Pain Episodes
Description: Assessed by using the Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-Me) Pain Episodes Short Form, which measures the frequency and severity of sickle cell pain episodes. 3 items are assessed using a scale that varies across the items, with values ranging from 0-7, 0-5, or 0-10, and the total raw score (minimum total score of 0 and maximum total score of 22) is rescaled into a standardized T-score. The standardized T-score has a mean of 50 and a standard deviation of 10. Higher T-scores indicate a worse outcome.
Time Frame: Baseline, week 4, week 8, and 4 weeks post-intervention (week 12)
Population: Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 19 | 25
T-score
  Baseline | 52.79 (7.66) | 45.84 (7.99)
  Week 4: number analyzed (Participants) | 11 | 23
  Week 4 | 49.32 (10.36) | 46.19 (9.72)
  Week 8: number analyzed (Participants) | 10 | 23
  Week 8 | 50.42 (9.01) | 44.87 (10.94)
  Week 12: number analyzed (Participants) | 10 | 19
  Week 12 | 48.55 (6.06) | 44.54 (8.51)

27. Secondary Outcome: Quality of Life: Emotional Impact
Description: Assessed by using the Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-Me) Emotional Impact Short Form, which measures the effects of sickle cell on emotional well-being. 5 items are assessed using a scale that ranges from 1 (always or very much) to 5 (never or not at all) and the total raw score (minimum total score of 5 and maximum total score of 25) is rescaled into a standardized T-score. The standardized T-score, with a minimum total score of 26.8 and a maximum total score of 65.6, has a mean of 50 and a standard deviation of 10. Higher T-scores indicate a better outcome.
Time Frame: Baseline, week 4, week 8, and 4 weeks post-intervention (week 12)
Population: Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 19 | 25
T-score
  Baseline | 51.70 (7.80) | 49.21 (6.45)
  Week 4: number analyzed (Participants) | 11 | 23
  Week 4 | 54.56 (8.54) | 52.57 (8.57)
  Week 8: number analyzed (Participants) | 10 | 23
  Week 8 | 55.13 (8.66) | 51.53 (8.98)
  Week 12: number analyzed (Participants) | 10 | 19
  Week 12 | 54.06 (6.92) | 52.84 (8.66)

28. Secondary Outcome: Quality of Life: Social Functioning
Description: Assessed by using the Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-Me) Social Functioning Short Form, which measures the influence of health on social functioning. 5 items are assessed using a scale that ranges from 1 (very much or always) to 5 (not at all or never) and the total raw score (minimum total score of 5 and maximum total score of 25) is rescaled into a standardized T-score. The standardized T-score, with a minimum total score of 26 and a maximum total score of 69.8, has a mean of 50 and a standard deviation of 10. Higher T-scores indicate a better outcome.
Time Frame: Baseline, week 4, week 8, and 4 weeks post-intervention (week 12)
Population: Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 19 | 25
T-score
  Baseline | 49.48 (10.52) | 51.43 (8.11)
  Week 4: number analyzed (Participants) | 11 | 23
  Week 4 | 56.04 (4.56) | 50.33 (8.08)
  Week 8: number analyzed (Participants) | 10 | 23
  Week 8 | 53.50 (8.34) | 51.92 (8.94)
  Week 12: number analyzed (Participants) | 10 | 19
  Week 12 | 57.82 (5.97) | 53.97 (10.58)

29. Secondary Outcome: Quality of Life: Stiffness Impact
Description: Assessed by using the Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-Me) Stiffness Impact Short Form, which measures joint/body stiffness. 5 items are assessed using a scale that ranges from 1 (always) to 5 (never) and the total raw score (minimum total score of 5 and maximum total score of 25) is rescaled into a standardized T-score. The standardized T-score, with a minimum total score of 24.9 and a maximum total score of 65.4, has a mean of 50 and a standard deviation of 10. Higher T-scores indicate a better outcome.
Time Frame: Baseline, week 4, week 8, and 4 weeks post-intervention (week 12)
Population: Participants who completed the corresponding survey for this outcome are included per timepoint.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | EaseVRx Group | Active Control Group
Number analyzed (Participants) | 19 | 25
T-score
  Baseline | 47.73 (6.62) | 45.78 (7.63)
  Week 4: number analyzed (Participants) | 11 | 23
  Week 4 | 52.20 (7.21) | 46.58 (6.13)
  Week 8: number analyzed (Participants) | 10 | 23
  Week 8 | 52.02 (7.76) | 47.06 (6.94)
  Week 12: number analyzed (Participants) | 10 | 19
  Week 12 | 54.78 (9.23) | 50.48 (7.56)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: The study involved a low-risk behavioral intervention for adults with SCD. An adverse event (AE) was considered as any event meeting the following definition:
  "Any untoward or unfavorable medical occurrence in a human subject, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the subject's participation in the research, whether or not considered related to the subject's participation in the research."
Arm/Group | EaseVRx Group | Active Control Group
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/25
Other Adverse Events (participants affected / at risk) | 1/19 | 0/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EaseVRx Group (N=19) | Active Control Group (N=25)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT04906707/Prot_SAP_001.pdf
  • Informed Consent Form (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT04906707/ICF_000.pdf